CLINICAL TRIAL: NCT06111118
Title: The Effectiveness of Sustained Heat Treatment on Delayed-Onset Muscle Soreness (DOMS) - An International, Multicenter, Open-label, Randomized Investigation
Brief Title: The Effectiveness of Sustained Heat Treatment on Delayed-Onset Muscle Soreness (DOMS)
Acronym: DOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 161(A)MD21047; 08600065397TC1FLX8000006U (Other: UNIQUE DEVICE IDENTIFICATION NUMBER); CIV-22-11-041492 (Other: german Ethic Commitee)
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Delayed-Onset Muscle Soreness (DOMS)
Keywords: HeatWraps Flexible; Thermacare; Medical Device; DOMS; Delayed-Onset Muscle Soreness; Heat therapy; Physical exercise
MeSH Terms: conditions — Hyperthermia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects who are qualified to enter the investigation will be randomized in a 2:2:1 ratio to one of the following 3 treatment groups, respectively:
  * Group 1: Immediate ThermaCare HeatWraps application (approximately 40 subjects)
  * Group 2: Delayed ThermaCare HeatWraps application (starting 24 hours after exercise; approximately 40 subjects)
  * Group 3: No treatment (approximately 20 subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate ThermaCare HeatWraps (Experimental): Immediately after the completion of standardized exercise ThermaCare HeatWraps will be applied on each leg centered over the quadriceps and lying longitudinally over the muscle for 8 hours. The application of a new ThermaCare HeatWraps will be repeated in the same manner, for 8 hours each, at 24 and 48 hours after exercise (i.e., 3 applications in total).
  Interventions: Device: ThermaCare HeatWraps
- Delayed ThermaCare HeatWraps (Experimental): On Day 2, 24 hours after the completion of standardized exercise, Group 2 subjects will apply ThermaCare HeatWraps in the same manner as described above for 8 hours. Subsequent heat wraps will be applied for 8 hours each at 48 and 72 hours after exercise (i.e., 3 applications in total).
  Interventions: Device: ThermaCare HeatWraps
- No treatment (No Intervention): Standardized exercise alone

INTERVENTIONS:
Device: ThermaCare HeatWraps — ThermaCare HeatWraps application
  Arms: Delayed ThermaCare HeatWraps; Immediate ThermaCare HeatWraps

SUMMARY:
This post-market clinical follow-up, open-label, multicenter, randomized, parallel group clinical investigation is designed to investigate the effectiveness, safety, and tolerability of immediate and delayed ThermaCare HeatWraps (medical device) applications against no treatment.

DETAILED DESCRIPTION:
This post-market clinical follow-up, open-label, multicenter, randomized, parallel group clinical investigation is designed to investigate the effectiveness, safety, and tolerability of immediate and delayed ThermaCare HeatWraps applications against no treatment.

Approximately 100 subjects, aged between 18 and 55 years (inclusive), will be enrolled into the investigation.

Having given informed consent and personal data processing consent, subjects will undergo a medical screening on Day 1 (Visit 1) to confirm their eligibility to enter the investigation.

Subjects who are qualified to enter the investigation will be randomized in a 2:2:1 ratio to one of the following 3 treatment groups, respectively:

* Group 1: Immediate ThermaCare HeatWraps application (approximately 40 subjects)
* Group 2: Delayed ThermaCare HeatWraps application (starting 24 hours after exercise; approximately 40 subjects)
* Group 3: No treatment (approximately 20 subjects) To induce DOMS, the subjects randomized into the investigation will perform a standardized exercise routine of squats between 14:00 and 15:00. An exercise monitor will set the pace at 3 seconds per squat, and subjects will be instructed to flex the hip past 110 degrees. Each set will last for 5 minutes followed by a 3-minute rest, which will be repeated two more times, for a total of 3 sets.

ELIGIBILITY:
Inclusion Criteria:

* Any gender and any ethnic origin, aged between 18 and 55 years (inclusive), in good general health and able to perform and complete the exercise regimen.
* No significant physical activity causing DOMS in the thighs/quads in the past 4 weeks.

Body mass index <40 kg/m2.

* No clinically relevant cardiovascular disease, hepatic disease, diabetes, lower limb neuropathies or recent lower limb injuries.
* Normal blood pressure (systolic blood pressure 90 to 140 mmHg, diastolic blood pressure 60 to 90 mmHg, inclusive) at rest.
* Subject is either not of childbearing potential (defined as biological male sex or postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) and must agree not to start a pregnancy from the signature of the informed consent up to the final visit or practicing one of the following medically acceptable methods of birth control:

  1. Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) up to the final visit
  2. Total abstinence from sexual intercourse since the last menses before exposure to the device and up to the final visit
  3. Intrauterine device
  4. Double-barrier method (condoms, sponge, diaphragm, with spermicidal jellies or cream) up to the final visit -----Must have personal smartphone (i.e., iOS or Android).
* Capable of returning to the investigation center for all the visits according to requirement of CIP.
* Willing to comply with the policy, procedure, and restriction of the investigation.
* Capable of actively communicating with the investigator.
* Capable of completing the investigation-related documents.
* Capable of understanding the contents of the informed consent and personal data processing consent and legally ---capable of signing a written informed consent and a personal data processing consent prior to any investigation-related procedures.

Exclusion Criteria:

* Skin lesions (e.g., rash, bruising, laceration) in the thigh region, or spreading skin conditions (e.g., poison ivy, urticaria) in other regions, or any skin abnormality likely to be aggravated by the device such as dermatological disease or infection, rash, atrophic, fragile or abnormally dry skin, cuts or abrasions at the treatment site.
* Clinically significant abnormalities at medical history and/or physical examination at Visit 1, which in the opinion of the investigator could interfere with the investigation procedures or endpoint evaluations.
* Treatment with alpha or beta agonists/antagonists, any type of anti-inflammatory or analgesic medications, Cox-2 inhibitors, calcium channel blockers, pregabalin (Lyrica), other pain reducers, muscle relaxants, creatine, ephedrine or pseudoephedrine.
* Lactating or pregnant women.
* Suspected or confirmed coronavirus disease 2019 infection at Visit 1.
* History of (within the past 12 months) or current alcohol or substance abuse.
* Any history of radiculopathy and neurological deficits.
* Vulnerable subjects (i.e., individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response).
* Subjects who have participated in another interventional investigation within the past 30 days before enrollment or are currently participating in another non-interventional investigation which might impact the outcome of this investigation.
* Subjects who are involved in the conduct of the investigation (i.e., investigator or his/her deputy, first grade relatives, pharmacist, assistant or other personnel).
* Known skin hypersensitivity to adhesion products.
* Any other condition that, in the opinion of the investigator, interferes with the investigation endpoints/procedures and does not justify the inclusion of the subject in the investigation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Difference in DOMS scores using an 11-point Numeric Rating Scale (NRS) | At 24 hours after exercise (Groups 1 and 3) and at 48 hours after exercise (Group 2)
  To assess the impact on DOMS pain through Numeric Rating Scale (NRS) after standardized exercise followed by an 8-hour ThermaCare HeatWraps application immediately following exercise or delayed application (24 hours after exercise) versus no treatment. The NRS is an 11-point scale scored from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable".

SECONDARY OUTCOMES:
Difference in DOMS scores using an 11-point Numeric Rating Scale (NRS) | at 8, 16, 48, and 72 hours after exercise (Groups 1 and 3) and at 32, 40, 72 and 96 hours after exercise (Group 2)
  Daily DOMS pain assessment through Numeric Rating Scale (NRS) across the duration of the entire investigation. The NRS is an 11-point scale scored from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable".
Subjects' global impression of perceived effect (muscle stiffness, ease of movement, flexibility, strength), therapeutic benefit and treatment satisfaction | At 8, 16, 24, 48 and 72 hours after exercise (Groups 1 and 3) and at 32, 40, 48, 72 and 96 hours after exercise (Group 2)
  Subjects' global impression of perceived effect through a unique Patient Global Impression of Severity (PGI-S) scale.
  The PGI-S is a 1-item questionnaire designed to assess subject's impression of DOMS severity. The subject will be asked to answer to the following questions:
  Based on your thigh's muscle soreness, how do you rate your muscle stiffness? Based on your thighs' muscle soreness, is there an impairment in your ease of movement? Based on your thighs' muscle soreness, is there an impairment in your flexibility? Based on your thighs' muscle soreness, is there any negative impact on your performance? Based on your thighs' muscle soreness, is there any negative impact on your muscle strength?
  The subject picks the answer that best describes his/her impression of DOMS severity, according to the PGI-S 7-point scale:
  1. Not present; 2.Very mild; 3. Mild; 4.Moderate; 5.Moderately severe; 6.Severe and 7. Extremely severe
Safety and Tolerability of ThermaCare HeatWraps | Through study completion, an average of 1 year
  Incidence of incidents/adverse events (AEs) as number of events

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - AMS Centro Médico del Ejercicio, Málaga, Malaga
  - Facultad Ciencias de la Salud Universidad de Malaga, Málaga, Malaga
  - Fisioterapia de la Serna, Madrid
  - Universidad Autonoma de Madrid (UAM) Hospital Universitario La Paz (HULP), Madrid
  - Medical Sportoledo, Toledo
  - Hospital Clinico Universitario de Valladolid, Valladolid